CLINICAL TRIAL: NCT00248586
Title: Development of Limited Contact CBT Treatment for IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03 DK67878 (completed 2007); R03DK067878 (NIH)
Record Dates: First submitted 2005-11-01; First posted 2005-11-04 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: IBS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard CBT (S-CBT) (Experimental)
  Interventions: Behavioral: Standard CBT (S-CBT)
- Minimal contact CBT (MC-CBT) (Experimental)
  Interventions: Behavioral: Minimal contact CBT (MC-CBT)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Standard CBT (S-CBT) — Standard CBT (S-CBT) is a skills-based training program delivered to patients in 10 weekly, 1-hour sessions.
  Arms: Standard CBT (S-CBT)
Behavioral: Minimal contact CBT (MC-CBT) — Minimal contact CBT (MC-CBT) covers the same range of procedures featured in S-CBT but relies extensively on self study materials.
  Arms: Minimal contact CBT (MC-CBT)

SUMMARY:
An accumulating body of evidence indicates that a specific psychological treatment called cognitive behavioral therapy (CBT) is associated with significant reductions in pain and bowel dysfunction of irritable bowel syndrome (IBS). Despite its apparent efficacy, the clinical effectiveness of CBT (i.e., its generalizability, feasibility, cost effectiveness) has not been adequately established due partly to its duration, cost, and limited accessibility. As the "second generation" of IBS treatments undergo development and validation, it has become increasingly clear that efficacy demonstration is a necessary but not sufficient condition of treatment viability. One potential solution to the problem of clinical effectiveness is to develop a briefer, largely self administered version of CBT that retains the efficacy of standard CBT but is more transportable, accessible, and less costly to deliver. To this end, a two-stage project is proposed. The goals of the first stage will be to develop, refine, and pilot test an innovative limited therapist contact-CBT protocol patterned after treatments proven effective for painful medical disorders with similar pathophysiology as IBS. The primary aim of the second stage is to conduct a small randomized clinical trial (N = 75 patients meeting Rome II diagnostic criteria) of standard (10 session) version of CBT (S-CBT) and limited contact (4 session) version of CBT (LC-CBT) with reference to a wait list control to examine their comparative efficacy on multiple indices, including IBS symptoms (primary outcome variable), psychological distress, and quality of life. Secondary aims are (1) to identify patient characteristics that predict outcome; (2) obtain information regarding active change-inducing mechanisms that may underlie treatment outcome; and (3) obtain information regarding possible monetary benefits, cost-effectiveness, and cost-benefit of S-CBT versus LC-CBT protocols. Data from this trial would set the stage for an R01 funded multicenter study with a large, random, and representative sample that could establish the clinical effectiveness of LC-CBT and in so doing make a significant contribution toward more efficient and effective care of IBS.

DETAILED DESCRIPTION:
An accumulating body of evidence indicates that a specific psychological treatment called cognitive behavioral therapy (CBT) is associated with significant reductions in pain and bowel dysfunction of irritable bowel syndrome (IBS). Despite its apparent efficacy, the clinical effectiveness of CBT (i.e., its generalizability, feasibility, cost effectiveness) has not been adequately established due partly to its duration, cost, and limited accessibility. As the "second generation" of IBS treatments undergo development and validation, it has become increasingly clear that efficacy demonstration is a necessary but not sufficient condition of treatment viability. One potential solution to the problem of clinical effectiveness is to develop a briefer, largely self administered version of CBT that retains the efficacy of standard CBT but is more transportable, accessible, and less costly to deliver. To this end, a two-stage project is proposed. The goals of the first stage will be to develop, refine, and pilot test an innovative limited therapist contact-CBT protocol patterned after treatments proven effective for painful medical disorders with similar pathophysiology as IBS. The primary aim of the second stage is to conduct a small randomized clinical trial (N = 75 patients meeting Rome II diagnostic criteria) of standard (10 session) version of CBT (S-CBT) and limited contact (4 session) version of CBT (LC-CBT) with reference to a wait list control to examine their comparative efficacy on multiple indices, including IBS symptoms (primary outcome variable), psychological distress, and quality of life. Secondary aims are (1) to identify patient characteristics that predict outcome; (2) obtain information regarding active change-inducing mechanisms that may underlie treatment outcome; and (3) obtain information regarding possible monetary benefits, cost-effectiveness, and cost-benefit of S-CBT versus LC-CBT protocols. Data from this trial would set the stage for an R01 funded multicenter study with a large, random, and representative sample that could establish the clinical effectiveness of LC-CBT and in so doing make a significant contribution toward more efficient and effective care of IBS.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria. To be included in the investigation, patients will have to: (a) be between the ages of 18 and 70 years of age; (b) meet Rome II criteria (66) for irritable bowel syndrome whose symptoms occur at least 2 days per week for 6 months or greater; (c) have a minimum 6th grade reading level based on the Wide Range Achievement Test (WRAT); (d) be willing to sign a consent form stating their willingness to participate in and participate in all phases of the investigation; (e) take either no IBS medications, or if taking medications, be on a stable dose for at least three months prior to trial entry with an understanding that dosage be maintained at pretreatment level(s) unless change is medically necessary.

Exclusion Criteria:

* Exclusion criteria. Patients will be excluded from the study if they (a) are undergoing concurrent psychological therapy and are unwilling or unable to stop treatment for the duration of the study; (b) have a history of having previously received actual CBT treatments being evaluated in the study, (c) have a diagnosed organic GI disorder or show current suicidality, substance abuse, psychosis in which case they will be referred for appropriate treatment; (e) are intellectually unable or unwilling to complete daily GI ratings

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Adequate relief - abdominal pain | 12 weeks
  In the past 7 days, have you had adequate relief from irritable bowel syndrome pain or discomfort?" (Yes/No).
Global symptom improvement | 12 weeks
  Compared to how you felt prior to entering the study, how would you rate the IBS symptoms for which you sought treatment during the past week?" (1, substantially improved; 4, no change; 7, substantially worse). Consistent with past research, we defined treatment responders a priori by a score of 1 (substantially) or 2 (moderately improved)

SECONDARY OUTCOMES:
IBS Quality of life | 12 weeks
Psychological distress | 12 weeks
  Global Severity Index of the Brief Symptom Inventory
IBS Symptom severity | 12 weeks
  IBS Symptom Severity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lackner, PsyD, Principal Investigator — UB, SUNY
Locations (1):
- UB, SUNY School of Medicine, Buffalo, New York, United States

REFERENCES:
- [Result] Lackner JM, Jaccard J, Krasner SS, Katz LA, Gudleski GD, Holroyd K. Self-administered cognitive behavior therapy for moderate to severe irritable bowel syndrome: clinical efficacy, tolerability, feasibility. Clin Gastroenterol Hepatol. 2008 Aug;6(8):899-906. doi: 10.1016/j.cgh.2008.03.004. Epub 2008 Jun 4. PMID 18524691
- [Derived] Lackner JM, Gudleski GD, Keefer L, Krasner SS, Powell C, Katz LA. Rapid response to cognitive behavior therapy predicts treatment outcome in patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2010 May;8(5):426-32. doi: 10.1016/j.cgh.2010.02.007. Epub 2010 Feb 17. PMID 20170751